CLINICAL TRIAL: NCT06234163
Title: The Effect of Enteral and Parenteral Nutrition Training Applied to Surgical Nurses on Their Knowledge Level and Care Behaviors Regarding Nutritional Care: Randomized Controlled Study
Brief Title: The Effect of Enteral and Parenteral Nutrition Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SINOPU-elif 1
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Enteral Nutrition; Parenteral Nutrition; Nursing Care
Keywords: EPN; Nutritional Care; Surgery; Care Behaviors
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention was made to the nurses in the control group (n = 35). In-service training is provided to nurses in this group in the clinic. After the study is completed, written material (brochure) was given to the nurses in the control group."Descriptive Survey Form" was applied at the beginning of the study. Other measurement tools, "Enteral and Parenteral Nutrition Care Knowledge Test" and "Care Behavior Scale-24 (BDI-24)" were applied three times as pre-test, post-test and follow-up test (three weeks later).
- Nutrition education group (Experimental): It was planned to give "Enteral and Parenteral Nutrition Training" to the nurses in the experimental group, based on the literature. The content of the training guide was sent to ten experts in the field and content validity was made. Enteral and parenteral nutrition training was given face to face, in 15-20 minutes, using verbal presentation and written materials (brochures). "Descriptive Survey Form" was applied to the experimental group (n=35) at the beginning of the research. Other measurement tools, "Enteral and Parenteral Nutrition Care Knowledge Test" and "Care Behavior Scale-24 (BDI-24)" were administered three times: before the training, within one or two days of the training and three weeks after the training.
  Interventions: Behavioral: Assigned intervention

INTERVENTIONS:
Behavioral: Assigned intervention — Enteral and parenteral nutrition training was given face to face, within 15-20 minutes, using oral presentation and written materials (brochures). The content of the "Enteral and Parenteral Nutrition Training Guide" prepared based on the literature was sent to ten experts in the field. and content validity was done. The training guide includes up-to-date information on topics such as enteral and parenteral nutrition indications and contraindications, evaluation of gastric residual volume, and nursing care in patients receiving enteral and parenteral nutrition.
  Other Names: Enteral and Parenteral Nutrition Training
  Arms: Nutrition education group

SUMMARY:
Malnutrition is considered as a deficiency of energy, protein or other nutrients. Malnutrition is a big problem for surgical patients. Various physiological problems may occur in patients with inadequate or malnutrition, such as prolonged wound healing time, decreased muscle strength and deterioration in immune system functions. It is recommended to start oral nutrition in the early postoperative period. In cases where the oral route is not preferred, enteral and parenteral nutritional support should be provided to the patient continuously or intermittently. Failure to identify individuals at risk of malnutrition means delaying the nutritional support the patient needs. Close observations and evaluations made by nurses during the day can ensure early diagnosis of the patient at risk of malnutrition and receive the necessary nutritional support. In order for nurses to fulfill their duties regarding nutritional care, they must have sufficient knowledge and skills on the subject and perceive the importance of nutritional care for patients. "Care" forms the basis of nursing. The interaction between patient and nurse affects the process and quality of care. Care behaviors include some basic skills such as listening carefully to the patient by making eye contact, empathy, demonsrating professional knowledge and skills, taking responsibility for the patient, and being accessible. In order to increase the quality of nursing care given to patients, it is necessary to provide evidence-based care and ensure that the care given is compatible with the values and expectations of the patients. For these reasons, this study aimed to examine the effect of enteral and parenteral nutrition (EPN) training on the knowledge level and care behaviors of surgical nurses regarding nutritional care.

DETAILED DESCRIPTION:
Sample Size and Statistical Methods:

The population of the research will consist of 199 nurses working in the surgical services and surgical intensive care units of Samsun 19 Mayıs University Faculty of Medicine Hospital between February 2024 and May 2024. The sample will consist of a total of 70 nurses (experiment = 35, control = 35) who meet the inclusion criteria for the study between the same dates. For the intervention and control groups; sampling criteria; Working as a nurse in a surgical ward or surgical intensive care unit and volunteering to participate in the study were defined as being eligible. Power analysis was performed to determine the number of people to be included in the study. The power of the test was calculated with the G*Power 3.1 program. As a similar study in the relevant literature, in the research conducted by Düdener (2019), the effect size regarding the difference in care behaviors was calculated as 0.647. In order to exceed the 95% value in determining the power of the study; At the 5% significance level and 0.615 effect size, 56 people, 28 people in the groups, need to be reached (df=27; t=1.703). In the research, it was aimed to reach a total of 70 people, 35 people in the groups, considering the high power of the test and the losses.

Nutrition Education Group

"Enteral and Parenteral Nutrition Training", prepared based on the literature, has been given to the nurses in the experimental group. The content of the training guide has been sent to ten experts in the field and content validity will be made. Enteral and parenteral nutrition training has been given face to face, in 15-20 minutes, using verbal presentation and written materials (brochures). "Descriptive Survey Form" will be applied to the experimental group (n=35) at the beginning of the research. Other measurement tools, "Enteral and Parenteral Nutrition Care Knowledge Test" and "Care Behavior Scale-24 (BDI-24)" hasbeen applied three times: before the training, within one or two days after the training and three weeks after the training.

Control group:

No intervention has been made to the nurses in the control group (n = 35). In-service training is provided to nurses in this group in the clinic. After the study is completed, written material (brochure) has been given to the nurses in the control group."Descriptive Survey Form" will be applied at the beginning of the study. Other measurement tools, "Enteral and Parenteral Nutrition Care Knowledge Test" and "Care Behavior Scale-24 (BDI-24)" has been applied three times as pre-test, post-test and follow-up test (three weeks later).

Data Collection Tools

"Descriptive Survey Form", "Care Behavior Scale-24 (BDI-24)" and "Knowledge Test on Enteral and Parenteral Nutritional Care" developed by the researchers were used to collect data in the study. The Knowledge Test on Enteral and Parenteral Nutritional Care was sent to ten experts along with the training guide to ensure content validity.

ELIGIBILITY:
Inclusion Criteria:

* Having the title of nurse
* Working in a surgical ward or surgical intensive care unit
* Volunteering to participate in the study

Exclusion Criteria:

• filling out forms incompletely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Knowledge Test on Enteral and Parenteral Nutritional Care | one day
  The "Knowledge Test on Enteral and Parenteral Nutritional Care (EPNB)" developed by the researchers consists of 45 items with "True" and "False" options. The content validity of the knowledge test will be carried out by ten experts in the field. In the EPNB Knowledge Test, 1 point is given for each correctly answered statement in the data set, and 0 point is given for each incorrectly answered statement. A minimum of 0 points and a maximum of 45 points in total can be obtained from the "EPNB Information Form".

SECONDARY OUTCOMES:
Care Behavior Scale-24 | one day
  Caring Behaviors Scale-24 (BDI-24) was created by Wu et al. (2006). The validity and reliability study of the scale was conducted by Kurşun and Kanan (2012) in our country. The scale was designed to evaluate the nursing care process. The scale is a six-point Likert type and consists of 24 items. The minimum total score obtained from the scale is 24 and the maximum is 144. Calculation of scale scores: Obtaining the total scale score: After adding the scores of 24 items, dividing by 24, a scale score between 1 and 6 is obtained. Obtaining sub-dimensions: For each sub-dimension, sub-dimension scores between 1-6 points are obtained by adding up the scores of the items in the sub-dimensions and dividing the resulting score by the number of items.

CONTACTS AND LOCATIONS:
Overall Officials: Sonay GÖKTAŞ, PhD, Study Director — Consulting
Locations (1):
- Elif ALTINKAYNAK SARAL, Sinop, Sinop University, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No